CLINICAL TRIAL: NCT07348445
Title: A Single-center, Randomized, Double-blind, Sham-controlled, Confirmatory Clinical Trial to Evaluate the Efficacy and Safety of the Digital Therapeutics (One.Dr) to Improve Blood Pressure Drop When Standing in Patients With Suspected Orthostatic Hypotension
Brief Title: Clinical Trial of Digital Therapeutics (One.Dr) for Suspected Orthostatic Hypotension Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1-2025-0056
Record Dates: First submitted 2026-01-09; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Hypotension; Orthostasis
MeSH Terms: conditions — Hypotension; Dizziness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One.Dr Application (Experimental)
  Interventions: Other: Digital therapeutics (One.Dr Application)
- Sham Application (Sham Comparator)
  Interventions: Other: Digital therapeutics (Sham Application)

INTERVENTIONS:
Other: Digital therapeutics (One.Dr Application) — An application that provides educations and non-pharmaceutical treatment (participant customized content) for orthostatic hypotension via a smart device
  Arms: One.Dr Application
Other: Digital therapeutics (Sham Application) — An application that provides general health knowledge via a smart device
  Arms: Sham Application

SUMMARY:
Participants who meet the inclusion/exclusion criteria in the Screening visit are randomly assigned 1:1 to the treatment group or the sham control group. The two-week period after Screening is the Run-in period, and the participant performs self-measured blood pressure monitoring, records data using the One.Dr application, and records symptoms and events related to orthostatic hypotension such as dizziness in the application. Only those who have completed the Run-in period will enter the Intervention period (for 6 weeks at 3-8 weeks), and according to each allocation group, non-pharmaceutical treatment education is provided for the treatment group and general health knowledge education is provided for the sham control group.

ELIGIBILITY:
Inclusion Criteria:

1. Adults over 19 years of age suspected of orthostatic hypotension due to symptoms such as dizziness within one year
2. Participants who are able to walk and conduct this clinical trial or cooperate with their care providers

Exclusion Criteria:

1. Participants diagnosed with diseases that cause dizziness other than orthostatic hypotension, such as otolithiasis and stroke, within one year
2. Severe anemia (Hb <8.0 g/dL, based on the latest test results within 12 months)
3. Participants unable to use smartphones (android phones) and/or smart watches
4. Participants with chronic diseases less than one year of life expectancy, such as malignant tumors
5. Participants with severe heart valve disease or severe heart failure (LVEF <35%) who have been hospitalized for acute exacerbation within the last 3 months
6. Participants with recent rapid and unintended weight loss (5% or more than 5 kg within 6 months)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
The changes in orthostatic SBP or DBP drop between the Run-in period and the Intervetion period | For 8 weeks after first use of digital therapeutics
  Orthostatic BP will be recorded during the Run-in period (2 wks) and the Intervetion period (6 wks). The orthostatic BP drops are expected to decrease in the treatment group than in the sham control group.

IPD SHARING:
Plan to Share IPD: Undecided